CLINICAL TRIAL: NCT07257692
Title: Reproducibility and Agreement of Appetite and Eating Behaviours in Response to Fixed Meals and the Modifying Effect of Feeding Status.
Brief Title: Effect of Feeding Status on Appetite and Eating Behaviour.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: University of Jazan (Other Government)
Responsible Party: Principal Investigator, James Dorling, PhD, Lecturer in Human Nutrition, Principal Investigator, University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 200220227
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eating behaviour trait questionnaires before the meal. (Other): Participants will complete the eating behaviour trait questionnaires before the meal.
  Interventions: Dietary Supplement: Standardised meal
- Eating behaviour trait questionnaires after the meal. (Other): Participants will complete the eating behaviour trait questionnaires after the meal.
  Interventions: Dietary Supplement: Standardised meal

INTERVENTIONS:
Dietary Supplement: Standardised meal — Participants will complete the wVAS (weekly visual analogue scale), the TFEQ (Three factor eating questionnaires)and the IES-2 (Intuitive eating scale-2)in the fasted state before the breakfast meal.
  Arms: Eating behaviour trait questionnaires before the meal.
Dietary Supplement: Standardised meal — Participants will be asked to complete the wVAS (weekly visual analogue scale), the TFEQ (Three factor eating questionnaires)and the IES-2 (Intuitive eating scale-2) 90 minutes after the administration of the breakfast meal.
  Arms: Eating behaviour trait questionnaires after the meal.

SUMMARY:
This clinical trial's primary aim is to evaluate the impact of a short-term feeding state on trait eating behaviours and weekly appetite. The secondary aim is to assess the relationship between appetite hormones (i.e., leptin, adiponectin, total glucagon-like peptide-1 (GLP-1), and peptide YY (PYY)) and long-term trait eating behaviours. The researchers will compare two groups (before vs. after a meal) to see if the meal affects appetite and eating behaviour traits in healthy adults.

DETAILED DESCRIPTION:
Study Design

Screening visit (Visit 1) Participants will be asked to complete a health screening questionnaire. Only those in generally good health will be enrolled. Following this, weight and height will be measured, and the body mass index (BMI) will be determined. Finally, participants will complete the International Physical Activity Questionnaire and food preferences questionnaire to ensure they like the foods provided in the study. Moreover, they will be provided with a 24-hour food diary to complete 24 hours before the first experimental trial, along with a set of scales to help them measure and record all items. Participants will be instructed to follow this food diary in the 24 hours before the second trial, ensuring that the food and drink consumed in the 24 hours before each experimental trial are similar.

Experimental trials (Visits 2 and 3) In the 24 hours prior to the experimental trial, participants will complete a 24-hour food diary where they record all food and beverages. With this diary, participants will describe all drinks and food consumed using household measures (e.g. teaspoon, cup). They will be asked to record a detailed description of food and/or drink intake, time and place of consumption. They will also record details on food brands, preparation and cooking methods. Portion sizes should be estimated using household measures or natural unit sizes (e.g., slices of bread). Food diaries and an electronic kitchen scale (Salter Housewares Ltd., Tonbridge, UK) will be provided to subjects, and they will be shown how to use the scales and how to record. They will follow this food diary in the 24 hours prior to the second visit to ensure they replicate their food and drink consumption in the 24 hours before each experimental trial.

Participants will arrive at the laboratory before both experimental trials at approximately 08:30, having fasted for at least 12 hours (participants instructed not to eat or drink after 20:30 from the previous night, except water). They will be weighed and then, at approximately 09:30, following a period of rest, a fasting blood sample will be collected by a researcher who is a trained phlebotomist. They will consume a standardised breakfast comprising porridge oats, full-fat milk, croissants, butter, jam and orange juice, which they will have 30 minutes to consume. Participants will then rest in the metabolic research unit for the remaining 3.5 hours of the trial (5-hour visit in total), completing study questionnaires where necessary. They will be able to consume water ad libitum and will be able to bring laptops/tablets and books.

During the experimental trial, participants will complete the weekly Visual Analogue Scale (wVAS), the Three Factor Eating Questionnaire (TFEQ) and the Intuitive Eating Scale-2 (IES-2) in the fasted state before the breakfast meal; while in the second trial, participants will be asked to complete these 90 minutes after the administration of the breakfast meal. In a randomised counter-balanced design, half of the participants will complete these scales in the fasted state first, whilst the other half will complete these scales after the breakfast meal first.

Throughout both experimental trials, participants will be periodically asked to complete measures of instantaneous appetite and food cravings. Instantaneous appetite ratings will be measured through the instantaneous Visual Analogue Scale (iVAS). These will examine various appetite constructs: hunger, satisfaction, fullness, prospective food consumption and desire to eat. Participants will be asked to place a vertical mark on the horizontal line at a point corresponding to their feelings at that time (hence the term instantaneous appetite). Participants will complete iVAS first at approximately 09:00, just before the breakfast meal. Thereafter, iVAS will be administered every 60 minutes (five assessments in total).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Have stable body mass for at least three months (within ±2 kg).

Exclusion Criteria:

* People who are younger than 18 or older than 65 years old.
* Have food allergies.
* SmokingTaking medications
* Suffering from metabolic health issues, e.g., history of diabetes, cardiovascular disease, or eating disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Dietary restraint | Once before the breakfast meal and once 90 minutes after the meal during each experimental trial.
  Dietary restraint is the cognitive effort or intention to consciously limit food intake of eating. Participants will complete assessments of the Three Factor Eating Questionnaire (TFEQ) (Stunkard et al., 1985) to assess restraint once at two different time points on each experimental trial in a randomised, counterbalanced fashion. The minimum score for restraint is 0 and the maximum is 20, with a higher score indicating higher levels of restraint.
Disinhibition | Once before the breakfast meal and once 90 minutes after the meal during each experimental trial.
  Disinhibition refers to the tendency to overeat in response to emotional, social, or situational cues, even when not physiologically hungry. Participants will complete assessments of the Three Factor Eating Questionnaire (TFEQ) (Stunkard et al., 1985) to assess disinhibition once at two different time points on each experimental trial in a randomised, counterbalanced fashion. The minimum score for disinhibition is 0, and the maximum is 16, with a higher score indicating greater disinhibition or loss of control over eating.
Hunger | Once before the breakfast meal and once 90 minutes after the meal during each experimental trial.
  Hunger reflects the subjective perception of appetite and the susceptibility to feelings of hunger and food cues. Participants will complete assessments of the Three Factor Eating Questionnaire (TFEQ) (Stunkard et al., 1985) to assess hunger once at two different time points on each experimental trial in a randomised, counterbalanced fashion. The minimum score for hunger is 0 and the maximum is 14, with a higher score indicating indicating greater susceptibility to feelings of hunger and greater responsiveness to food cues.
Unconditional Permission to Eat (UPE) | Once before the breakfast meal and once 90 minutes after the meal during each experimental trial.
  Unconditional Permission to Eat reflects a person's ability to allow themselves to eat a wide range of foods without guilt or unnecessary rules. It captures how flexible and trusting someone is toward their own hunger cues. Participants will complete the Intuitive Eating Scale-2 (IES-2) (Tylka & Kroon Van Diest, 2013) to assess UPE at two time points during each experimental trial in a randomised, counterbalanced order. Items are rated on a 5-point scale from 1 (strongly disagree) to 5 (strongly agree), with higher scores indicating a greater ability to permit oneself to eat when hungry without external restrictions.
Eating for Physical Rather Than Emotional Reasons (EPR) | Once before the breakfast meal and once 90 minutes after the meal during each experimental trial.
  Eating for Physical Rather Than Emotional Reasons reflects the extent to which individuals eat in response to genuine physical hunger rather than emotions such as stress, boredom, or sadness. This construct captures a healthy separation between emotional states and eating behaviour. Participants will complete the IES-2 (Tylka & Kroon Van Diest, 2013) at two time points during each experimental visit in a randomised, counterbalanced order. Items are scored on a 1-5 scale, with higher values indicating a stronger tendency to eat based on physical hunger rather than emotional triggers.
Reliance on Hunger and Satiety Cues (RHSC) | Once before the breakfast meal and once 90 minutes after the meal during each experimental trial.
  Reliance on Hunger and Satiety Cues measures how effectively individuals listen to and trust their internal bodily signals to guide when, what, and how much to eat. It reflects a mindful and attuned approach to eating. Participants will complete the IES-2 (Tylka & Kroon Van Diest, 2013) at two different time points on each study day in a randomised, counterbalanced fashion. Items are rated on a 5-point scale, and higher scores indicate stronger trust in one's internal cues of hunger and fullness.
Body-Food Choice Congruence (BFCC) | Once before the breakfast meal and once 90 minutes after the meal during each experimental trial.
  Body-Food Choice Congruence reflects how consistently individuals choose foods that support their physical functioning, health, and well-being. It captures a compassionate connection between how a person feels and the types of foods they select. Participants will complete the IES-2 (Tylka & Kroon Van Diest, 2013) at two time points during each experimental visit in a randomised, counterbalanced design. Items use a 1-5 response scale, with higher scores indicating greater alignment between food choices and physical self-care.
Hunger | Once before the breakfast meal and once 90 minutes after the meal during each experimental trial.
  Hunger represents how frequently and intensely participants felt hungry over the past week. Using the weekly Visual Analogue Scale (wVAS) (Womble et al., 2003), participants rate their overall hunger on a 100-mm line from 0 mm (not hungry at all during the week) to 100 mm (extremely hungry throughout the week). Higher scores indicate stronger or more frequent hunger sensations during the previous week.
Fullness | Once before the breakfast meal and once 90 minutes after the meal during each experimental trial.
  Fullness reflects how often or how strongly participants felt full across the previous week. Using the weekly Visual Analogue Scale (wVAS) (Womble et al., 2003), participants will complete the wVAS, marking fullness on a 100-mm scale from 0 mm (rarely or never felt full during the week) to 100 mm (felt very full very often throughout the week). Higher scores indicate more frequent or stronger feelings of fullness across the week.
Satisfaction | Once before the breakfast meal and once 90 minutes after the meal during each experimental trial.
  Satisfaction reflects how content or pleased participants felt with their eating experiences during the past week. Using the weekly Visual Analogue Scale (wVAS) (Womble et al., 2003), participants rate satisfaction on a 0-100 mm line from 0 mm (not satisfied at all during the week) to 100 mm (extremely satisfied with eating throughout the week). Higher scores indicate greater overall satisfaction during the week.
Desire to Eat | Once before the breakfast meal and once 90 minutes after the meal during each experimental trial.
  Desire to eat reflects how frequently participants experienced an urge or motivation to eat during the previous week. Using the weekly Visual Analogue Scale (wVAS) (Womble et al., 2003), participants will rate this on the wVAS, from 0 mm (little or no desire to eat during the week) to 100 mm (strong desire to eat very often throughout the week). Higher scores indicate a stronger or more frequent desire to eat during the past week.

SECONDARY OUTCOMES:
Plasma Leptin Concentration | Before breakfast meal (fasting state).
  A single fasting blood sample to measure the circulating levels of leptin (ng/mL) concentration, measured using ELISA.
Plasma Adiponectin Concentration | Before breakfast meal (fasting state).
  A single fasting blood sample to measure the circulating levels of adiponectin (µg/mL) concentration, measured using ELISA.
Plasma Glucagon-Like Peptide-1 (GLP-1) Concentration | Before breakfast meal (fasting state).
  A single fasting blood sample to measure the circulating levels of GLP-1(pmol/L) concentration, measured using ELISA.
Plasma Peptide YY (PYY) Concentration | Before breakfast meal (fasting state).
  A single fasting blood sample to measure the circulating levels of PYY (pg/mL) concentration, measured using ELISA.
Plasma Gastric Inhibitory Polypeptide (GIP) Concentration | Before breakfast meal (fasting state).
  A single fasting blood sample to measure the circulating levels of GIP (pg/mL) concentration, measured using ELISA.
Plasma C-Reactive Protein (CRP) Concentration | Before breakfast meal (fasting state).
  A single fasting blood sample to measure the circulating levels of CRP (mg/L) concentration, measured using ELISA.
Plasma Insulin Concentration | Before breakfast meal (fasting state).
  A single fasting blood sample to measure the circulating levels of Insulin (µU/mL) concentration, measured using ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: James Dorling, PhD, Principal Investigator — University of Glasgow
Locations (1):
- New Lister Building at Glasgow Royal Infirmary, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The stored data will be anonymous and follow the guidelines of the General Data Protection Regulation enforced in May 2018. Hard copies of participant information forms, including consent forms and dietary intake records, will be kept in locked filing cabinets. Keys to the filing cabinets will only be available to the primary investigator. All databases will be password protected and stored on a university computer with firewalls.
  Participants' identifiable data will be stored in a locked cabinet. Digital data will be stored anonymously within the server of the University of Glasgow.
  This project's Principal Investigator will be responsible for sharing the research data.
  Data will be preserved in Enlighten, the official online repository of Glasgow University's research output.
Time Frame: The data will be available when the study is completed. Data will be preserved for 10 years.
Access Criteria: Data will be shared via the repository deposit (Enlighten). Only signatories of end-user agreements can access and use shared data.

REFERENCES:
- [Background] Stunkard AJ, Messick S. The three-factor eating questionnaire to measure dietary restraint, disinhibition and hunger. J Psychosom Res. 1985;29(1):71-83. doi: 10.1016/0022-3999(85)90010-8. PMID 3981480
- [Background] Tylka TL, Kroon Van Diest AM. The Intuitive Eating Scale-2: item refinement and psychometric evaluation with college women and men. J Couns Psychol. 2013 Jan;60(1):137-53. doi: 10.1037/a0030893. PMID 23356469
- [Background] Womble LG, Wadden TA, Chandler JM, Martin AR. Agreement between weekly vs. daily assessment of appetite. Appetite. 2003 Apr;40(2):131-5. doi: 10.1016/s0195-6663(02)00170-8. PMID 12781162